CLINICAL TRIAL: NCT01180907
Title: The Biodistribution of 1-[2 Deoxy-2, -18 Fluroarabinfuranosyl]Cytosine [18FAC] in Healthy Subjects and Patients With Cancer, Autoimmune/Inflammatory Diseases: A Pilot Study
Brief Title: The Biodistribution of 1-[2 Deoxy-2, -18 Fluroarabinfuranosyl]Cytosine [18FAC] in Healthy Subjects and Patients With Cancer, Autoimmune/Inflammatory Diseases
Status: Completed | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 07-07-071; DE-PS02-08ER-08-01 (Other Grant/Funding Number: Department of Energy); CIRMNo. RT1-01126-1 (Other Grant/Funding Number: California Institute for Regenerative Medicine); 10-000269 (Other: UCLA Medical IRB#2)
Record Dates: First submitted 2010-08-11; First posted 2010-08-12 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Cancer; Inflammation
Keywords: 18F-FAC; imaging; cancer; inflammation; PET
MeSH Terms: conditions — Neoplasms; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- patients with cancer
- patients with autoimmune diseases
- healthy subjects

SUMMARY:
The purpose of the study is to determine whether positron emission tomography using the new imaging agent 18F-FAC can be used for imaging cancer and/or inflammation.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* women of childbearing potential will undergo a pregnancy test free of charge
* patients with cancer or autoimmune diseases or healthy subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with cancer, autoimmune diseases and healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-11; Primary Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christiaan Schiepers, M.D. Ph.D, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States